CLINICAL TRIAL: NCT04431375
Title: Efficacy of Addition of Fecal Microbiota Transplant (FMT) and Plasma Exchange to Tenofovir in Comparison to Monotherapy With Tenofovir in ACLF-HBV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-05
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Acute-On-Chronic Liver Failure; Hepatitis B
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis B | interventions — Plasma Exchange; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plasma Exchange+Tenofovir+FMT (Experimental): Subjects will receive Plasma exchange 2 sessions alternate day followed by FMT for 7 days and Tenofovir [antiviral] 300mg PO once a day .
  Interventions: Biological: Plasma Exchange; Drug: Tenofovir; Other: Fecal Mircobiota Transplantation
- Tenofovir (Active Comparator): TabletTenofovir [antiviral] 300mg per oral once a day
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Biological: Plasma Exchange — Plasma exchange 2 sessions alternate day followed by FMT for 7 days and Tenofovir [antiviral] 300mg PO once a day .
  Arms: plasma Exchange+Tenofovir+FMT
Drug: Tenofovir — Tenofovir [antiviral] 300mg PO once a day .
Other: Fecal Mircobiota Transplantation — FMT for 7 days
  Arms: plasma Exchange+Tenofovir+FMT

SUMMARY:
A randomized controlled trial to study the efficacy of addition of FMT & plasma exchange to tenofovir compared to monotherapy with tenofovir in patients with HBV reactivation who develops Acute on chronic liver failure.

In this study the patients who meet the inclusion criteria will be randomized to either receive Tenofovir or with FMT + plasma exchange along with Tenofovir . Blood samples & stool samples will be taken & analysis will be done accordingly .The patients are followed for 90 days MELD,APACHE & SOFA scores are calculated.Then statistical analysis will be done to find whether the addition of plasma exchange & FMT adds benefit compared to tenofovir treatment alone .

DETAILED DESCRIPTION:
A randomized controlled trial to study the efficacy of addition of FMT & plasma exchange to tenofovir compared to monotherapy with tenofovir in patients with HBV reactivation who develops Acute on chronic liver failure.

In this study the patients who meet the inclusion criteria will be randomized to either receive Tenofovir or with FMT + plasma exchange along with Tenofovir . Blood samples & stool samples will be taken & analysis will be done accordingly .The patients are followed for 90 days MELD,APACHE & SOFA scores are calculated.Then statistical analysis will be done to find whether the addition of plasma exchange & FMT adds benefit compared to tenofovir treatment alone .

Study period: 2 Years

Intervention:

The patients in Group A will receive T.Tenofovir [antiviral] 300mg per oral once a day .

The patients in Group B will receive Plasma exchange 2 sessions alternate day followed by FMT for 7 days and Tenofovir [antiviral] 300mg PO once a day .

Intravenous antibiotics will be given to all patients included in study empirically, because of high risk of infection in these patients. Patients with sepsis are excluded from the study.

Methodology for FMT - Fresh Stool [30 g] is obtained from donor <3 hr before FMT. 150 mL sterile 0.9N saline is added to sample & homogenized in a blender. It is Continued 3 times in pulses of 20-30 secs, till homogenous suspension. Slow filtration is done with membrane filter (330µm) to give adequate time. Filtration is repeated 3 times. Patient is kept NPO for 4 hrs. prior to the instillation .100 ml of fresh filtrate is given for 7 days through naso-jejunal tube over 5-10 minutes .Patient is kept reclined at 45° for 4 hr. Normal diet is given after 2 hr of procedure. IV antibiotics are continued as per institutional protocol in case of sepsis.

Methodology for plasma exchange [PE] - Circulatory access will be established through a double lumen catheter via the patient's femoral vein. The total exchanged plasma volume will be 2500-3500 mL, and the Plasma Exchange rate will be 20-25 mL/min. Fresh-frozen plasma (FFP) will be supplied by the ILBS Blood Bank. Dexamethasone (5 mg) and heparin (2500 U) will be injected routinely before PE. Heparin will be neutralized at the end of PE by an injection of 20-50 mg protamine sulfate. PE will be repeated alternate day for a total of 2 sessions Adverse effects: FMT FMT - Sore throat and difficulty in deglutition secondary to naso-gastric tube insertion Plasma exchange PE

* Hypocalcemia
* Hypokalemia
* Metabolic alkalosis
* Hypotension
* Anaphylaxis
* TRALI TENOFOVIR Tenofovir
* Reversible proximal renal tubular toxicity.
* Reduced bone mineral density
* Manifestations of mitochondrial toxicity (i.e., neuropathy, myopathy, lactic acidosis

Stopping rule of study:

* Allergic reactions except mild drug reactions
* Arterial hypotension or development of shock /Hypertension
* Arrhythmias
* Development or progression of organ failures during therapy
* Transfusion related lung injury
* Uncontrolled Bleeding or DIC
* Severe dyselectrolytemia( k+<2.5 or >5.5)
* Seizures/tetany
* Patients who are undergoing or listed for Transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age - 18-75 years
* Patients with ACLF - HBV reactivation according to APASL guidelines.
* MELD < 30 WITH AKI,HE
* MELD < 30 WITH OUT EXTRAHEPATIC FAILURE

Exclusion Criteria:

* MELD > 30
* Co existing hepatitis A,E,D
* HCC
* Sepsis
* Alcohol intake, substance abuse, HIV, IBD, chronic constipation or diarrhoea
* Allergy to plasma, protamine or heparin,
* Active hemorrhage or disseminated intravascular coagulation (DIC)
* Unstable hemodynamics (e.g., blood pressure <90/60 mmHg, heart rate >100 bpm),
* Cerebral or myocardiac infarction
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival in both groups | Day 28

SECONDARY OUTCOMES:
Overall survival in both groups | 3 months
Reduction in HBV DNA level | 14 days
Reduction in HBV DNA level | 60 days
Reduction in HBV DNA level | 90 days
Reduction in CTP Score in both groups | 14 days
  CTP Score ranges from 5 to 15 5=good 15=worst
Reduction in CTP Score in both groups | 30 days
  CTP Score ranges from 5 to 15 5=good 15=worst
Reduction in CTP Score in both groups | 60 days
  CTP Score ranges from 5 to 15 5=good 15=worst
Reduction in CTP Score in both groups | 90 days
  CTP Score ranges from 5 to 15 5=good 15=worst
Reduction in MELD Score in both groups | 14 days
  MELD Score ranges from 6 to 40 6=good 40=worst
Reduction in MELD Score in both groups | 30 days
  MELD Score ranges from 6 to 40 6=good 40=worst
Reduction in MELD Score in both groups | 60 days
  MELD Score ranges from 6 to 40 6=good 40=worst
Reduction in MELD Score in both groups | 90 days
  MELD Score ranges from 6 to 40 6=good 40=worst
Percentage of patient's with improvement in hepatic failure calculated by MELD Na and CTP scores. | 14 days
Percentage of patient's with improvement in hepatic failure calculated by MELD Na | 30 days
Percentage of patient's with improvement in hepatic failure calculated by CTP scores. | 30 days
Percentage of patient's with improvement in hepatic failure calculated by MELD Na | 60 days
Percentage of patient's with improvement in hepatic failure calculated by CTP scores. | 60 days
Percentage of patient's with improvement in hepatic failure calculated by MELD Na. | 90 days
Percentage of patient's with improvement in hepatic failure calculated by CTP scores. | 90 days
Change in microbiota profile in both groups | 10 days
Change in microbiota profile in both groups | 30 days
Change in microbiota profile in both groups | 60 days
Change in microbiota profile in both groups | 90 days
Change in plasma cytokine profile in both groups | 10 days
Change in plasma cytokine profile in both groups | 28 days
Change in plasma cytokine profile in both groups | 60 days
Number of patients with adverse Events in both groups | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided